CLINICAL TRIAL: NCT00269503
Title: A Pilot Study of Chiropractic Prone Distraction for Subacute Back Pain With Sciatica
Brief Title: Chiropractic Prone Distraction for Lower Back Pain
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Samueli Institute for Information Biology (Other)
Collaborators: National Naval Medical Center (U.S. Federal Agency)
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: #B04-091
Record Dates: First submitted 2005-12-21; First posted 2005-12-23 (Estimated); Last update posted 2008-05-08 (Estimated); Status verified 2008-05

CONDITIONS: Herniated Disc; Lower Back Pain; Sciatica
MeSH Terms: conditions — Intervertebral Disc Displacement; Low Back Pain; Sciatica | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant

INTERVENTIONS:
Procedure: Prone Distraction
Procedure: Side-Posture Manipulation
Procedure: Side-Posture Manipulation & Prone Distraction
Procedure: Usual Care (Control Group)

SUMMARY:
Back pain is a major cause of disability in the United States. The lifetime prevalence of low back pain is estimated at 60-90%. Back pain has conservatively been estimated to involve total direct and indirect costs of over $25 billion annually in lost wages, treatment, and related issues. These losses clearly extend to the active duty population cared for by military health care facilities.

Chiropractic medicine is characterized by the use of a number of physical manipulations and mobilization techniques, which can be used singly or in combination to treat a variety of medical conditions. Although basic clinical practice guidelines for Chiropractic have been developed, few studies have rigorously compared techniques and their outcomes for specific conditions. Fewer still have sought to correlate treatment modality with both anatomical effect and clinical outcome.

Throughout the military, Chiropractic care is available only to active duty personnel and only at a limited number of medical treatment facilities. At National Naval Medical Center, it is a well-established treatment option, where the full array of techniques is employed, primarily for painful conditions, and most often for back pain. This study seeks to clarify the mechanisms of action and efficacy of one specific treatment option, prone distraction, for the relief of subacute sciatica due to radiographically confirmed herniated disc, and to compare it to side-posture manipulation and standard medical management.

Prone lumbar distraction utilizes a specialized table with motorized continual motion distraction. This table has multiple mechanical articulations that can be used to place patients in a wide variety of positions. Patients being treated with continuous motion distraction are placed prone with the table positioned for maximum comfort and centralization of symptoms.

Side posture manipulation is a widely practiced, standard chiropractic technique, which has been shown to provide considerable clinical improvement for patients with sciatica. Low- grade oscillatory stresses are performed within the physiological range of normal joint motion. The hip, pelvis and lumbar spine are rotated forward with manual pressure while a counter rotation of the chest and thoracic spine is applied.

ELIGIBILITY:
Inclusion Criteria:

* Active Duty military personnel
* Aged 18-45 (age is limited to 45 years due to the natural aging and degeneration of the discs; the less hydration the disc maintain, the less likely manipulation will be successful).
* Have subacute low back pain (more than three months duration but less than six months duration), with radicular component (sciatica) rated at a minimum level of 4 on the Numerical Rating Scale (NRS) of the Brief Pain Inventory
* Have a confirmed herniated disc, as noted on MRI, which correlates with the clinical findings (sciatica)

In this study, a "herniated disc" refers to any localized displacement of disc material, including nucleus, cartilage, fragmented apophyseal bone, or fragmented anular tissue, which results in back and leg pain. "Herniated Disc" also will include disc extrusions and disc bulges (protrusions) only when with associated annular tears.

In this study, "sciatica" refers to pain in the lower extremity/ies that follows the course of the sciatic nerve

Exclusion Criteria:

* Patients who are not able to give informed consent.
* Pregnant or nursing women
* Patients who have a primary bone disease, cancer, infection, spondylolysis or spondylolisthesis.
* Patients who have had prior spine surgery, including rhizotomy
* Participation in another conflicting research study
* Patients who cannot commit to a trial lasting up to eight weeks or cannot come for bi-weekly treatments
* Patients who are going through a course of physical therapy or chiropractic treatment or at the time of planned enrollment or are being currently being managed and/or treated for any pain condition
* Patients who have an unstable medical or psychiatric condition
* Patients who are planning or have been advised to have spine surgery
* Any contraindications to either prone distraction or side posture manipulation will disqualify potential subjects from any participation in this study
* Patients with a pacemaker.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2006-03; Primary Completion 2006-06 (Actual); Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
Change in overall leg pain intensity, as assessed by the change, if any, of leg pain documented on the Numerical Rating Scale (NRS) in the Brief Pain Inventory (BPI) from baseline to 8 weeks
Time to pain relief, defined as NRS less than 4 after 2 consecutive visits

SECONDARY OUTCOMES:
Change in overall back pain intensity, as assessed by the change, if any, of back pain documented on the BPI from baseline to 8 weeks
Change in overall pain intensity, as assessed by the change, if any, of the sum of back and leg pain documented on the BPI at measured intervals
Change in overall pain intensity, as assessed by the change, if any, of the sum of back and leg pain documented on the BPI from baseline to 8 weeks
Patient satisfaction with treatment, as assessed by The Client Satisfaction Questionnaire
Medication use, as assessed by the Medication Log
Functional disability, as assessed by The Roland-Morris Low Back Pain and Disability Questionnaire
Lost/decreased workdays
Change, if any, in percent of disc herniation, as determined by the study neuroradiologist
Descriptive changes in disc morphology, as assessed by the study neuroradiologist
Variability of treatment, as assessed by the number or prescriptions written, the number of visits to the Primary Care Clinic, as well as the number of referrals to additional treatments outside of the chiropractic clinic

CONTACTS AND LOCATIONS:
Overall Officials: William E Morgan, DC, Principal Investigator — National Naval Medical Center; CDR Robert E Rosenbaum, MC, USN, Principal Investigator — National Naval Medical Center
Locations (1):
- National Naval Medical Center, Bethesda, Maryland, United States